CLINICAL TRIAL: NCT00493675
Title: Biodegradable Biliary Stent for Post Operative Cystic Duct Leakage. Pilot Study
Brief Title: Biodegradable Biliary Stent for Post Operative Cystic Duct Leakage
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulties in getting suitable applicators for biodegradable stents.
Sponsor: Tampere University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R06089
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-02

CONDITIONS: Cyst
Keywords: Cystic duct leakage
MeSH Terms: conditions — Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: endoscopic bile duct stenting

SUMMARY:
Endoscopic sphincterotomy and temporary stenting is a routine treatment for post cholecystectomy cystic duct leakage. The draw back is that the plastic stent need to be removed later in a second intervention. Our studies with animal models have demonstrated that biodegradable biliary stent is at least as good as conventional plastic stent to heal that kind of leakage. In this pilot study the biodegradable biliary stent is inserted endoscopically to patients with confirmed cystic duct leakage to demonstrate the efficacy in human setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed post cholecystectomy cystic duct leakage requiring endoscopic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Clinical healing of bile leakage | 1 month

SECONDARY OUTCOMES:
Laboratory tests for liver function, ultra sound for bile collections and bile duct diameter and abdominal plain X-ray for stent degradation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Juhani A Sand, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland